CLINICAL TRIAL: NCT05291143
Title: The Effectiveness of Short Videos on Knowledge of Proper Home Blood Pressure Monitoring (HBPM) Among Malaysian Medical Students
Brief Title: The Effectiveness of Short Videos on HBPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Aneesa Abdul Rashid, Family Medicine Specialist and medical lecturer, Universiti Putra Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UPMG112022
Record Dates: First submitted 2022-03-10; First posted 2022-03-22 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Hypertension; Blood Pressure
Keywords: hypertension; blood pressure; home monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: educational video
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): This arm will get the educational video intervention
  Interventions: Behavioral: Short videos on blood pressure monitoring

INTERVENTIONS:
Behavioral: Short videos on blood pressure monitoring — Short videos on blood pressure monitoring

SUMMARY:
Hypertension prevalence among Malaysian adults is high at around 30% and is also reported to be the highest risk factor for mortality in Malaysia. Home Blood Pressure Monitoring (HBPM) has been proven to improve blood pressure levels for at least twelve months when used in conjuction with co-inventions such as education interventions or support from health care professionals. Social media has been described as having a favourable role in health interventions due to its popularity with vast numbers of users particularly the younger adults, its advantages mainly in health communication with patients, plus its promising impact on behavioural change. It has been reported that around 15% of those with hypertension are young adults; aged between 18-39 years. Therefore, this may be a good start to plan an intervention program on hypertension using the concept of short videos as popularised by social media; particularly on home blood pressure monitoring. As students are future doctors and can act as advocate in sharing important healthcare knowledge to family members and friends, they are the best candidate to be chosen as subjects of this research.

DETAILED DESCRIPTION:
Background

Hypertension is a major global public health problem, affecting about 1.13 billion people worldwide. It is often poorly controlled leading to many health complications, particularly cardiovascular diseases. Patients with hypertension are often managed in the primary care setting, where the use of home blood pressure monitoring (HBPM) is an effective tool for diagnosing and managing hypertension. HBPM has been proven to improve blood pressure levels for at least twelve months when used in conjunction with co-inventions such as education interventions or support from health care professionals.

Around 15% of those with hypertension are young adults; aged between 18-39 years. The definition of 'young hypertension', however, has been defined as up to 45 years old. Developing hypertension at a young age puts this group at risk of earlier onset cardiovascular events. Nonetheless, there are many challenges in treating hypertension in young adults, including the perception that it is a disorder for older people; lack of health education; shortage of suitable educational materials; and limited health resources.

In order to engage with this group, social media has been described as having a favourable role in health interventions due to its popularity with vast numbers of users particularly the younger adults, its advantages mainly in health communication with patients, plus its promising impact on behavioural change.

In Malaysia, internet use is 88.7% in 2020, and 70.5% use internet at home making Malaysia's access to the internet higher than the world's average, however a little lower than the UK levels at around 94.6%. Internet accessibility is also available to the rural population as shared by a study done in the state of Sabah. As many as 93.3% use internet for social media with Facebook and WhatsApp being the most popular applications used. It is apparent that the young adults from the age range 20-49 makes up the majority of internet users. In the UK, it has been reported that those aged between 25-34 makes up for the largest group on Facebook.

Systematic reviews have reported social media as a good communication tool assisting target users on a variety of health-related conditions. Some studies have shown positive change in behaviours affecting weight loss, fitness, sexual health and smoking cessation but citing limitation such as heterogenicity in meta-analysis and suggestions for better intervention designs. There are other concerns with regards to social media use like the spread of inaccurate, unregulated and harmful information, privacy issues, besides the exposure to harmful behaviours for example cyberbullying. Nevertheless, it may hold valuable potential in helping practitioners with the management of hypertension as social media could lead to better knowledge and awareness on the condition, assist in decision making and increase in health related self-efficacy. Therefore, suggesting the need for trusted resources from social media platforms, that health care professionals can use to signpost to, especially for the younger patients.

Hence, with findings of large studies, along with expert recommendations on the effectiveness of hypertension management with a HBPM program with co-inventions, social media may have a promising impact as a support tool specifically those in the younger age group to better manage their condition. The development of a social media assisted HBPM program will also help in future works for healthcare providers who may want to adopt this effort.

Problem Statement It has been reported that around 15% of those with hypertension are young adults; aged between 18-39 years. In order to engage with this group, social media has been described as having a favourable role in health interventions due to its popularity among this age group. Therefore, this may be a good start to plan an intervention program on hypertension using the concept of short videos as popularised by social media; particularly on home blood pressure monitoring. As students are future doctors and can act as advocates in sharing important healthcare knowledge to family members and friends, they are the best candidate to be chosen as subjects of this research.

Significance of Study Hypertension is a major global public health problem and around 15% of those with hypertension are young adults. The use of home blood pressure monitoring (HBPM) is an effective tool for diagnosing and managing hypertension. Therefore knowledge on HBPM is essential. Using an intervention program on hypertension using the concept of short videos as popularised by social media can be a good way to teach students on its concept. Hence, this study will determine the effectiveness of this mode of presentation to teach young adults on HBPM. This concept may later be extended to the public

Objectives General To determine the effectiveness of short videos on knowledge on HBPM among medical students Specific

1. To identify the socio-demographic data of students in this study
2. To determine the level of knowledge on HBPM pre intervention (short video)
3. To determine the level of knowledge on HBPM post intervention (short video).
4. To determine the effectiveness of HBPM short videos on knowledge of HBPM among medical students

Study Hypothesis The HBPM short video is effective in increasing knowledge on HBPM

Methodology Study Location: Faculty of Medicine and Health Sciences, UPM Study Design: This pre-post cross sectional study is conducted over a period of 3 months during the research module for undergraduate students their level of knowledge will be assessed pre, post watching the video and 2 weeks after. No control group is included due to resource constraints.

Study Duration:

Sampling Study population All year 2 UPM medical students

Sampling frame A list of year 2 medical students obtained from the Deputy Dean (Academic: Medical) office Sampling unit A year 2 medical student

Sampling method Universal sampling

Sample size All year 2 medical students will be approached to participate in the study. The estimated number of students are around 100 students Tools for assessment Study instrument on social media use was adapted from a previously published questionnaire which was a study about Health Information Seeking and Social Media Use on the Internet among people with Diabetes[20]. The questionnaire on HBPM was developed from literature review and consists of 20. Validation of this section will be done using content validation.

Face validation for all the questions will be done with 10% of the sample size and content validation will be done with expert panel consisting of family medicine specialists, public health medicine specialists and internal medicine specialists.

The questionnaire will be in 3 sections:

1. Sociodemographic factors Students' age, gender, ethnicity, religion, family monthly income and length of internet use. There is a total of 6 questions.
2. Social media use questionnaire The respondents were assessed the type of social media use and rate the duration of different types of social media used with 14 questions. The respondents were allowed to choose if they use social media daily or number of times a week, they use social media. The respondents were also allowed to state their average hours per day of using social media
3. HBPM There will be 20 questions on BP monitoring. All questions are based on the latest Malaysian Hypertension CPG. Respondents may pick either yes or no as the answer. Each correct question warrants 1 point. The higher the marks, the better the knowledge

Intervention:

There are 3 videos around 1 minute on important information on HBPM 1st video: 4 things you need to avoid 30 minutes before measuring your blood pressure (8) 2nd video How to take a proper home blood pressure measurement (8) 3rd video How to take accurate blood pressure measurement (8)

Data collection Data will be collected using an online questionnaire. This will be disseminated email. Reminders will be sent every week to remind participants to answer.

Data Analysis The data will be analysed using IBM Social Package for Social Science (SPSS) version 26 (30). In descriptive analysis, we will determine frequency and percentage for categorical data. Continuous data will be tested for normality using Kolmogorov-Smirnov and Shapiro-Wilk statistics and graphically using histogram, stem-and-leaf plots, and normal probability plot and detrended normal plots. If the data is normally distributed, mean, and standard deviation will be reported in the result but if the data is not normally distributed, we will use the median and interquartile range. The associations between the level of knowledge with other factors, respectively will be determined using the multiple linear regression modelling. Factors at univariate analysis of p value <0.200 will be included the model to determine these associations. All hypothesis testing will apply 2-sided test with level of significance at p= 0.05.

Research Ethics This study's approval for ethical clearance will be obtained from Medical Research Ethics Committee University Putra Malaysia (JKEUPM). Informed consent will be obtained from each study participant, and they will be told the right not to respond to the questions they don't want to respond or to terminate the online questionnaire at any time. If they agree to participate, they need to sign the e-consent form with digital signature. All data obtained will be kept confidentially and for research purposes only.

Variables Dependent variables The level of knowledge on HBPM

Independent variables

1. Socio-demographic factors Age Sex Religion Ethnicity

Expected Outcomes knowledge score pre and post intervention

ELIGIBILITY:
Inclusion Criteria:

* All year 2 medical students in UPM

Exclusion Criteria:

* Students who are acutely ill during the study period

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
knowledge score on home blood pressure monitoring (HBPM) | 3 months
  knowledge score is used to asses the level of HBPM knowledge. minimum score is 0, maximumum score is 20. The higher the score, the better the knowledge
knowledge score on home blood pressure monitoring (HBPM) | 12 months
  knowledge score is used to asses the level of HBPM knowledge. minimum score is 0, maximumum score is 20. The higher the score, the better the knowledge

CONTACTS AND LOCATIONS:
Overall Officials: Aneesa Abdul rashid, MBBCh BAO, Principal Investigator — Universiti Putra Malaysia
Locations (1):
- Universiti Putra Malaysia, Seri Kembangan, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
All data and materials analysed may be accessed if deemed appropriate by contacting the principal investigator

REFERENCES:
- [Result] Rashid AA, Ghazali SS, Mohamad I, Mawardi M, Musa H, Roslan D. The effectiveness of a Malaysian House Officer (HO) preparatory course for medical graduates on self-perceived confidence and readiness: A quasi-experimental study. PLoS One. 2020 Jul 17;15(7):e0235685. doi: 10.1371/journal.pone.0235685. eCollection 2020. PMID 32678838
- [Result] McManus RJ, Mant J, Franssen M, Nickless A, Schwartz C, Hodgkinson J, Bradburn P, Farmer A, Grant S, Greenfield SM, Heneghan C, Jowett S, Martin U, Milner S, Monahan M, Mort S, Ogburn E, Perera-Salazar R, Shah SA, Yu LM, Tarassenko L, Hobbs FDR; TASMINH4 investigators. Efficacy of self-monitored blood pressure, with or without telemonitoring, for titration of antihypertensive medication (TASMINH4): an unmasked randomised controlled trial. Lancet. 2018 Mar 10;391(10124):949-959. doi: 10.1016/S0140-6736(18)30309-X. Epub 2018 Feb 27. PMID 29499873
- [Result] Schwartz JE, Muntner P, Kronish IM, Burg MM, Pickering TG, Bigger JT, Shimbo D. Reliability of Office, Home, and Ambulatory Blood Pressure Measurements and Correlation With Left Ventricular Mass. J Am Coll Cardiol. 2020 Dec 22;76(25):2911-2922. doi: 10.1016/j.jacc.2020.10.039. PMID 33334418